CLINICAL TRIAL: NCT05909995
Title: A Phase 1 Study of INCB099280 in Combination With Ipilimumab in Participants With Select Solid Tumors
Brief Title: Interventional Study of INCB 99280 With Ipilimumab in Participants With Select Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a strategic business decision. There were no safety concerns contributing to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 99280-205; 2023-503243-34-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Melanoma; Hepatocellular Carcinoma (HCC); Renal Cell Carcinoma (RCC); Microsatellite Instability - High (MSI-H); Mismatch Repair Deficient (dMMR); Colorectal Carcinoma (CRC)
MeSH Terms: conditions — Melanoma; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Turcot syndrome; Colorectal Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): * Participants with RCC and MSI-H/dMMR CRC will receive 1 of two doses of INCB099280 BID with up to 4 doses of ipilimumab 1 mg/kg Q3 weeks
  * Participants with Melanoma and HCC will receive 1 of 2 doses of INCB099280 BID with up to 4 doses of 3 ipilimumab 3 mg/kg Q3 weeks
  Interventions: Drug: INCB 99280 with Ipilimumab
- Dose Expansion (Experimental): * Participants with RCC will receive 1 of two doses of INCB099280 BID with up to 4 doses of ipilimumab 1 mg/kg Q3 weeks of ipilimumab
  * Participants with HCC will receive 1 of two doses of INCB099280 BID with up to 4 doses of ipilimumab 3 mg/kg Q3 weeks of ipilimumab
  Interventions: Drug: INCB 99280 with Ipilimumab

INTERVENTIONS:
Drug: INCB 99280 with Ipilimumab — Dose Escalation and expansion of INCB 99280 with Ipilimumab

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, PK, and efficacy of INCB 99280 in combination with ipilimumab in participants with select solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Prior systemic therapy, diagnoses and disease setting as follows:

  * For Part 1 (dose escalation), and no history of treatment with anti-CTLA-4 or anti-PD-(L)1 therapy and one of the following,

    * Unresectable or metastatic cutaneous melanoma, or
    * Unresectable of metastatic Child-Pugh Class A NDD not eligible for surgical and/or locoregional therapy, or
    * Intermediate or poor-risk advanced clear cell RCC, or
    * MSI-H or dMMR metastatic CRC and able to provide fresh or archival tumor tissue for central confirmation of MSI-H or dMMR.
  * For Part 2 (dose expansion), IO treatment -naïve, e.g., no prior receipt of an anti PD-1, anti-PD-L1 or PD-L1, anti-CTLA-4, GITR, LAG3, TIM3, OX-40, IL-2, 4-1BB or other immune modulator, and have not received prior systemic therapy and one of the following,

    * Unresectable or metastatic Child-Pugh Class A HCC not eligible for surgical and/or locoregional therapy, or
    * Intermediate - or poor-risk advanced clear cell RCC.
  * ECOG performance score of 0 or 1.
  * Life expectancy > 3 months, in the opinion of the investigator.
  * Histologically confirmed solid tumors with measurable disease per RECIST v1.1.

    * Exception: HCC may be diagnoses based on cross-sectional multiphasic imagining using the AASLD criteria.
  * Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Known history of an additional malignancy.
* Central nervous system (CNS) metastases requiring treatment and/or leptomeningeal disease.
* Toxicity from prior therapy that has not recovered.
* Received thoracic radiation within 6 months of the first dose of study treatment.
* Participation in another interventional clinical study while receiving INCB099280.
* Impaired cardiac function of clinically significant cardiac disease.
* History of evidence of interstitial lung disease including non-infections pneumonitis.
* Presence of gastrointestinal condition that may affect drug absorption
* Any autoimmune disease requiring systemic treatment in the past 5 years.
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy at a daily dose exceeding 10 mg of prednisone or equivalent
* Active infection requiring systemic therapy.
* History of organ transplantation, including allogeneic stem cell transplantation.
* Receipt of system antibiotics within 28 days of first dose of study treatment.
* Probiotic usage is prohibited during the screening and throughout the study treatment period.
* Received a live vaccine within 28 days of planned start of study drug.
* Laboratory values outside the Protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Occurence of DLTs | 2 Years
Incidence of TEAEs | 2 Years
  Assessed by physical examinations, changes in vital signs and ECGs, and analysis of clinical laboratory samples.
Incidence of TEAEs leading to dose interruption, dose reduction, or discontinuation of either of the study drugs | 2 Years

SECONDARY OUTCOMES:
Concentration of INCB099280 in plasma | 2 Years
Objective response | 2 Years
  Defined as having a best overall response of complete response or partial response by investigator assessment per RECIST v1.1.
Disease control | 2 Years
  Defined as having a best overall response of complete response or partial response, or stable disease of ≥ 15 weeks after initiation of study treatment, by investigator assessment per RECIST v1.1.
Duration of Response | 2 Years
  Defined as the time from the earliest date of CR or PR until the earliest date of disease progression (by investigator assessment per RECIST v1.1) or death due to any cause if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Valkyrie Clinical Trials, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Henry Ford Health System, Detroit, Michigan
  - Alliance For Multispecialty Research Llc, Knoxville, Tennessee
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- South Africa (2):
  - Johese Clinical Research: Midstream, Centurion
  - Mary Potter Oncology Centre, Pretoria